CLINICAL TRIAL: NCT01215838
Title: Dynamic Contrast Evaluation of the Liver Using Gadoxetate Disodium (Eovist®) for Hepatocellular Carcinoma (HCC)
Brief Title: MRI of the Liver With Eovist
Status: Terminated | Type: Observational
Why Stopped: Unable to meet enrollment expectations.
Sponsor: University of Washington (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: DI-2009-1; 7160 (Other: FHCRC)
Record Dates: First submitted 2010-09-28; First posted 2010-10-07 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; hepatocellular carcinoma; Eovist; MR; MRI; magnetic resonance
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if a new magnetic resonance (MR) protocol is better at diagnosing liver lesions.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC), a form of liver cancer, is the seventh most common cause of cancer mortality in the US. The incidence rate of HCC is increasing along with the incidence of Hepatitis B and C which are known to promote HCC. Patients have a better prognosis (survival outlook) if HCC is found and treated at an early stage. MRI is the best imaging modality for diagnosing HCC.

This study will compare standard MRIs and MRIs performed with a newly developed MR protocol to determine if it is possible to more confidently diagnose HCC.

ELIGIBILITY:
Inclusion Criteria:

* known hepatocellular carcinoma
* undergoing MRI of the liver

Exclusion Criteria:

* Contraindication to MRI with IV contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known hepatocellular carcinoma undergoing MRI of the liver in the UWMC Radiology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of a new MR protocol in diagnosing HCC and other liver lesions. | One day: participants will have one MRI of the liver.

CONTACTS AND LOCATIONS:
Overall Officials: Orpheus Kolokythas, MD, Principal Investigator — University of Washington

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Background] Saito K, Kotake F, Ito N, Ozuki T, Mikami R, Abe K, Shimazaki Y. Gd-EOB-DTPA enhanced MRI for hepatocellular carcinoma: quantitative evaluation of tumor enhancement in hepatobiliary phase. Magn Reson Med Sci. 2005;4(1):1-9. doi: 10.2463/mrms.4.1. PMID 16127248
- [Background] Frericks BB, Loddenkemper C, Huppertz A, Valdeig S, Stroux A, Seja M, Wolf KJ, Albrecht T. Qualitative and quantitative evaluation of hepatocellular carcinoma and cirrhotic liver enhancement using Gd-EOB-DTPA. AJR Am J Roentgenol. 2009 Oct;193(4):1053-60. doi: 10.2214/AJR.08.1946. PMID 19770329